CLINICAL TRIAL: NCT07323498
Title: Enhancing Generalization of Virtual Reality Exposure for Public Speaking Anxiety Via Imagery-Based Extinction Memory Updating: A Randomized Controlled Trial
Brief Title: Enhancing Generalization of Virtual Reality Exposure for Public Speaking Anxiety
Acronym: VREX2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Christoph Benke, Principal Investigator, Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VREX2.0
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Public Speaking Anxiety; Public Speaking Fear
Keywords: virtual reality exposure; extinction generalization; fear extinction; exposure therapy
MeSH Terms: conditions — Glossophobia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR Exposure + Standard Mental Rehearsal (Active Comparator): Single-session VR exposure intervention: 6 VR speech exposure trials & Post-exposure standard mental rehearsal
  Interventions: Behavioral: VR Exposure; Behavioral: Standard Mental Rehearsal
- VR Exposure + Mental Rehearsal With Extinction Memory Updating (Experimental): Single-session VR exposure intervention: 6 VR speech exposure trials & Post-exposure mental rehearsal with updating the extinction memory with novel, non-exposed contexts
  Interventions: Behavioral: VR Exposure; Behavioral: Mental Rehearsal With Extinction Memory Updating

INTERVENTIONS:
Behavioral: VR Exposure — 6 VR speech exposure trials (3 min each; topic: "something you are proud of")
Behavioral: Standard Mental Rehearsal — Post-exposure guided imagery: vivid mental rehearsal of the same exposure experience in the same VR contexts (brief, ≤30s each)
  Arms: VR Exposure + Standard Mental Rehearsal
Behavioral: Mental Rehearsal With Extinction Memory Updating — Post-exposure guided imagery: vivid rehearsal of the exposure experience while updating the extinction memory with novel, non-exposed contexts (e.g., speaking to three real listeners; speaking in a new VR context with a larger audience). Brief, ≤30s each
  Arms: VR Exposure + Mental Rehearsal With Extinction Memory Updating

SUMMARY:
This randomized controlled trial examines whether imagery-based extinction memory updating following a standardized virtual reality (VR) exposure session improves the generalization of exposure effects to novel public speaking contexts. Individuals with elevated public speaking anxiety will complete a single-session VR speech exposure. Participants are randomized to (a) standard mental rehearsal of the exposure experience or (b) mental rehearsal plus guided imagery that updates the extinction memory with novel, non-exposed contexts. Generalization is assessed 7-14 days later using a multi-context behavioral approach test (BAT) in vivo and in VR.

DETAILED DESCRIPTION:
Exposure-based interventions are highly effective in the treatment of anxiety disorders; however, fear reduction achieved during exposure is often limited to the specific situations and stimuli encountered during treatment. As a result, fear may re-emerge when individuals face novel situations, a phenomenon commonly referred to as return of fear. This limited generalization is assumed to reflect the context- and stimulus-specific nature of extinction learning. While increasing variability across exposure contexts can enhance generalization, this approach typically requires longer treatment duration and increased therapeutic burden. Therefore, strategies that promote extinction generalization without increasing exposure time are of high clinical relevance.

Experimental laboratory research has demonstrated that extinction generalization can be enhanced by updating the extinction memory through mental imagery. Specifically, retrieving a recently acquired extinction memory and integrating novel, non-experienced stimuli or situations through imagination has been shown to reduce fear responses to both imagined and previously unencountered stimuli. This process is thought to increase the accessibility and robustness of inhibitory extinction memories by integrating new information into the existing memory network. The present study aims to translate this experimentally established mechanism into a clinically relevant intervention.

In this randomized controlled trial, individuals with elevated public speaking anxiety complete a standardized, single-session virtual reality (VR) speech exposure consisting of repeated short oral presentations across different VR contexts. Following exposure, participants are randomized to one of two imagery-based post-exposure procedures. In the control condition, participants engage in guided mental rehearsal of the previously experienced VR exposure situations. In the experimental condition, participants additionally update the extinction memory by vividly imagining having the same successful exposure experience in two novel public speaking situations: (1) giving a speech in front of a small real audience and (2) giving a speech in a VR environment with a substantially larger audience than experienced during exposure. These imagined situations are not directly experienced during the intervention but are intended to be integrated into the existing extinction memory through guided imagery.

Generalization of exposure effects is assessed 7-14 days after the intervention using a multi-context behavioral approach test (BAT). The BAT includes oral presentations in (a) situations that were directly experienced during VR exposure, (b) situations that were previously imagined during the extinction memory updating procedure, and (c) novel situations that were neither experienced nor imagined before. This design allows for the differentiation between responses to previously experienced, imagined, and entirely new public speaking contexts, thereby providing a stringent test of extinction generalization.

Primary outcomes include public speaking anxiety at follow-up as well as subjective fear ratings during each behavioral approach test, with a focus on differences between study groups across the different BAT contexts. Secondary outcomes include anticipatory anxiety prior to each BAT and behavioral performance indexed by speech duration. Baseline measures of anhedonia and positive emotionality are assessed to examine individual differences in treatment response.

ELIGIBILITY:
Inclusion Criteria:

* speech anxiety scale score of ≥ 18 on the Personal Report of Communication Apprehension, Public Speaking Subscale (PRCA-PS)
* Self-report of 18 - 70 years of age

Exclusion Criteria:

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-11-26 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Public Speaking Anxiety | From enrollment to one-week follow-up assessment
  Assessed using the Personal Report of Communication Apprehension, Public Speaking Subscale (PRCA-PS). Scores range from 6 to 30, with higher scores associated with higher public speaking anxiety.
Subjective Fear During Behavioral Approach Tests | one-week follow-up assessment
  Self-reported fear during oral presentations, rated on a scale from 0 (no fear) to 100 (severe fear) during each behavioral approach test. Participants were instructed to speak for up to three minutes and could terminate the task at any time.
  BAT 1: Oral presentation in vivo in front of 3 real listeners BAT 2: Oral presentation in a simulated videoconference with a large audience (30 listeners) BAT 3: Oral presentation in virtual reality (exposure context 1; familiar) BAT 4: Oral presentation in virtual reality (exposure context 2; familiar) BAT 5: Oral presentation in virtual reality (novel context with ~50 virtual listeners) BAT 6: Oral presentation in virtual reality (novel context with ~100 virtual listeners)

SECONDARY OUTCOMES:
Social Anxiety Severity | From enrollment to one-week follow-up assessment
  Severity of social anxiety symptoms assessed using the Social Phobia Inventory (SPIN). Scores range from 0-68, with higher scores indicating greater social phobia.
Anticipatory Anxiety Before BATs | One-week follow-up assessment
  Self-reported anticipatory anxiety assessed immediately before each behavioral approach test on a scale from 0 (no fear) to 100 (severe fear).
Behavioral Performance During BATs (Duration of oral presentation during BATs) | One-week follow-up assessment
  Duration of oral presentation during each behavioral approach test, measured in seconds. Participants were instructed to speak for up to three minutes and could terminate the task at any time.
Valence of Public Speaking | From enrollment to immediately post-treatment assessment and one-week follow-up assessment
  Self-report measure assessing how participants feel about having to give a speech. Valence is rated on a 7-point Likert scale ranging from extremely unpleasant to extremely pleasant (-3 = extremely unpleasant, -2 = moderately unpleasant, -1= slightly unpleasant, 0 = neutral, 1= slightly pleasant, 2= moderately pleasant, 3=extremely pleasant). Higher scores indicate more pronounced pleasantness.
Anticipated Fear of Public Speaking | From enrollment to immediately post-intervention and 1-week follow-up
  Participants rate their anticipated fear of giving a speech using a visual analog scale ranging from 0 (no fear) to 100 (extreme fear).

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Benke, Ph.D., Principal Investigator — Philiips-University of Marburg
Locations (1):
- Department of Psychology, Philipps-University of Marburg, Marburg, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No